CLINICAL TRIAL: NCT02162849
Title: The Effects of Behavioral Counseling Plus Nicotine Replacement Therapy (NRT) or Varenicline on Smoking Cessation Among Smokers High and Low in Intrinsic Reward Sensitivity
Brief Title: Reward Sensitivity and Pharmacotherapy for Smoking Cessation
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: NAL PHARMA (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-0207; NCI-2014-01485 (Registry Identifier: NCI CTRP); RP140262 (Other Grant/Funding Number: CPRIT)
Record Dates: First submitted 2014-06-11; First posted 2014-06-13 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Tobacco Use Cessation
Keywords: Tobacco Use Cessation; Smoking Cessation; Cancer Prevention; Behavioral Counseling; Nicotine Replacement Therapy; NRT; Nicotine patch; Placebo patch; Placebo pill; Sugar pill; Varenicline; Chantix; Questionnaires; Surveys; Saliva test
MeSH Terms: conditions — Tobacco Use Cessation; Smoking Cessation | interventions — Varenicline; Tobacco Use Cessation Devices; Sugars; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Varenicline + Placebo Patch (Experimental): Varenicline dosing follows the recommended 12 week course: 0.5 milligram mg/day by mouth for Days 1-3, 0.5 mg twice a day for Days 4-7, and 1 mg twice a day thereafter. Participant takes Varenicline 1-10 days after Visit 1.
  Starting on Day 8, and then every day after that, participant applies 1 placebo patch each day.
  Questionnaire completion 1 to 10 days before first study drug/placebo dose and on Days 8, 17, 24, 31, 38, 52, and 73. On Days 17, 24, 38, and 73, done over the phone.
  Counseling sessions performed on Days 8, 17, 24, 31, 38, 52, and 73. On Days 17, 24, 38, and 73, done over the phone. During counseling on Day 8, participant sets a "quit date" for stopping smoking for about 1 week after participant starts taking the study drug/placebo. Some of the counseling sessions may be recorded by video and/or audio tape.
  Study staff calls participant 1 day before quit date and 3 days after quit date to check on progress in quitting smoking.
  Interventions: Drug: Varenicline; Drug: Placebo Patch; Behavioral: Questionnaires; Behavioral: Counseling Sessions; Other: Lab Session; Other: Saliva Test
- Nicotine Patch + Placebo Tablet (Experimental): Participant takes placebo tablet 1-10 days after Visit 1. On Days 1-3, participant takes 1 dose of the placebo each morning. Starting on Day 4, and then every day after that, participant takes 1 dose in the morning and 1 dose in the evening.
  Starting on Day 8, and then every day after that, participant applies 1 nicotine patch.
  Questionnaire completion 1 to 10 days before first study drug/placebo dose and on Days 8, 17, 24, 31, 38, 52, and 73. On Days 17, 24, 38, and 73, done over the phone.
  Counseling sessions performed on Days 8, 17, 24, 31, 38, 52, and 73. On Days 17, 24, 38, and 73, done over the phone. During counseling on Day 8, participant sets a "quit date" for stopping smoking for about 1 week after participant starts taking the study drug/placebo.
  Study staff calls participant 1 day before quit date and 3 days after quit date to check on progress in quitting smoking.
  Interventions: Drug: Nicotine Patch; Drug: Placebo Tablet; Behavioral: Questionnaires; Behavioral: Counseling Sessions; Other: Lab Session; Other: Saliva Test

INTERVENTIONS:
Drug: Varenicline — Varenicline Dosing: 0.5 mg/day by mouth for Days 1-3; 0.5 mg twice a day for Days 4-7, and 1 mg twice a day thereafter.
  Other Names: Chantix
  Arms: Varenicline + Placebo Patch
Drug: Nicotine Patch — Starting on Day 8, and then every day after that, participant applies 1, 21 mg nicotine patch for 11 weeks.
  Arms: Nicotine Patch + Placebo Tablet
Drug: Placebo Patch — Starting on Day 8, and then every day after that, participant applies 1 placebo patch each day for 11 weeks.
  Arms: Varenicline + Placebo Patch
Drug: Placebo Tablet — Participant takes placebo tablet 1-10 days after Visit 1. On Days 1-3, participant takes 1 dose of the placebo each morning. Starting on Day 4, and then every day after that, participant takes 1 dose in the morning and 1 dose in the evening.
  Other Names: Sugar pill
  Arms: Nicotine Patch + Placebo Tablet
Behavioral: Questionnaires — Questionnaire completion 1 to 10 days before first study drug/placebo dose and on Days 8, 17, 24, 31, 38, 52, and 73. Questionnaires should take about 30-45 minutes total to complete. On Days 17, 24, 38, and 73, done over the phone.
  Other Names: Surveys
Behavioral: Counseling Sessions — Counseling sessions performed on Days 8, 17, 24, 31, 38, 52, and 73. On Days 17, 24, 38, and 73, done over the phone. These sessions take about 15 minutes each time.
Other: Lab Session — Participant asked to watch slides. During the lab session, brain electrical activity checked with an electroencephalogram (EEG). Participant completes computer tasks, including questionnaires, that will measure emotions and attention level. These tasks should take about 90 minutes to complete. The lab session may last up to 2 hours.
Other: Saliva Test — Saliva tested to check cotinine level at baseline, on Days 8 and 17, end of treatment visit, and at 3 months and 6 months after quitting smoking.

SUMMARY:
The goal of this clinical research study is learn if varenicline or the nicotine patch can help people with different types of emotion and attention levels to quit smoking.

DETAILED DESCRIPTION:
Study Groups:

If you agree to take part in this study, you will be randomly assigned (as in the roll of a dice) to 1 of 2 study groups. This is done because no one knows if one study group is better, the same, or worse than the other group. You will have an equal chance of being assigned to Group 1 or 2.

* If you are in Group 1, you will receive varenicline and a placebo patch. A placebo is not a drug. It looks like the study drug but is not designed to treat any disease or illness. It is designed to be compared with a study drug to learn if the study drug has any real effect.
* If you are in Group 2, you will receive an active nicotine patch and a placebo tablet.

Neither you nor the study doctor will know which group you are assigned to. However, if needed for your safety, the study staff will be able to find out what you are receiving (called "unblinding").

Once the study has ended and the Data Safety Monitoring Board (DSMB) at MD Anderson has granted approval, you may be unblinded at your request.

Study Drug Administration:

You will start taking your assigned study drug(s) the day after Visit 1.

You should take varenicline/placebo tablets by mouth with a cup (8 ounces) of water after eating a full meal. On Days 1-3, you will take 1 dose of the study drug each morning. Starting on Day 4, and then every day after that, you will take 1 dose in the morning and 1 dose in the evening (for a total of 2 doses of the study drug each day). You must return any study drug bottles as well as any unused study drug to the study staff at each study visit.

You should apply the nicotine/placebo patch to the upper arm. You should put it in a slightly different place each day to avoid skin irritation. You may take the patch off at night to avoid sleeping problems.

You will be given a study diary to record how many cigarettes you smoke (if any) each day while you are on study.

You must return your study diary and any unused study drugs, patches, and/or containers at each study visit.

Study Visits (Visits 1-7):

At every study visit:

* You will complete questionnaires about several topics, including depression, suicide, your smoking behavior, and any effects from the study drug. These questionnaires should take about 30-45 minutes in total to complete.
* You will be giving the opportunity to complete the questionnaires verbally with a study staff member (either on phone or in person depending on the visit number) or electronically on your computer using a website administered by an online survey development company called Qualtrics.
* You will receive counseling about quitting smoking, where you will talk about possible "triggers" for smoking and strategies for dealing with quitting smoking. These sessions will take about 15 minutes each.

At Visits 1, 4 and 6:

* Urine or saliva will be collected for a routine test to check your cotinine, nicotine, and anabasine levels. Cotinine is a chemical released in your body when it breaks down nicotine and will show whether and how much you have recently smoked. Anabasine is used to show if nicotine is found in the blood due to a nicotine replacement therapy or from tobacco use.
* Your CO level and weight. will be measured.
* If you did not have one during screening, you will have a physical exam.
* If you did not complete at one during screening or before Visit 1, you will complete the EEG/lab session.
* If you can become pregnant, urine will be collected for a pregnancy test.
* At V1, if your CO machine tests results are unclear, and the study staff thinks it is appropriate, a NicAlert test will be performed. Urine will be collected for the NicAlert test, which is more sensitive at detecting levels of smoking than the CO machine.

During counseling on Day 8, you will set a "quit date" for stopping smoking for about 1 week after you start taking the study drug/placebo. You should not quit smoking before the quit date. You may also set goals to reduce smoking. You should try to stay smoke-free after the quit date. You will also be given a drug instruction sheet, a card with emergency contact information, and a participant manual to help you follow along with the topics discussed during counseling.

Visits 2, 3, 5 and 7 will be conducted over the phone. You will complete questionnaires about several topics (either on the phone or electronically), including depression, mood, your smoking behavior, and any effects from the study drug. You will also be asked about any drugs you may be taking. Each call should take about 25-45 minutes.

The study staff will call you 1 day before your quit date and 3 days after your quit date to check on your progress in quitting smoking. Each call should take about 10-15 minutes.

Lab Session:

You will take part in a lab session at or before Visit 1 to test your brain activity. You will be asked to watch slides. The slides will include pictures of people, nature, and artwork. Slides showing nude people, medical procedures, and victims of car crashes will also be shown. You will be shown examples of these slides before beginning the procedure and given the opportunity to withdraw from the study.

During the lab session, your brain electrical activity will be checked with an electroencephalogram (EEG). To do this, small sensors will be placed on your scalp and face. You should not drink more than 2 cups of coffee or other caffeinated drinks for at least 2½ hours before the session. At the lab session, you may be asked to smoke a cigarette if the doctor thinks it is needed for you to show your normal smoking behavior.

You will also complete computer tasks, including questionnaires that will measure your emotions and attention level. These tasks should take about 90 minutes to complete.

The lab session may last up to 2 hours.

Ecological Momentary Assessments (EMA):

EMA are used to gather information about your mood and cravings as they happen in your day-to-day life. At your randomization visit, you will be loaned a smart phone device, and will be asked to complete questionnaires on the device at different times everyday throughout the active treatment phase (12 weeks). In these questionnaires, you will be asked about events from the previous day, such as cigarettes per day, alcohol intake, mood, sleep, motivation, and whether you took your prescribed drugs on time. These questionnaires should take up to about 20 minutes per day to complete.

Length of Treatment:

You will receive the study drug/placebo for up to 12 weeks. You will be taken off study early if the doctor thinks it is in your best interest or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visits.

End-of-Treatment Visit (Visit 8):

After you have finished taking the study drug/placebo, the following tests and procedures will be performed:

* Your CO level will be measured.
* Blood (about 2 teaspoons) will be drawn to check your liver and kidney function.
* Urine or saliva will be collected to measure your nicotine, anabasine, and cotinine level.
* You will complete the same questionnaires you completed at the regular study visits.
* You will receive counseling about quitting smoking.
* If you can become pregnant, urine will be collected for a pregnancy test.

Follow-Up Visits (Visits 9 and 10):

At about 3 and 6 months after you have stopped smoking, the following tests and procedures will be performed:

* Your CO level will be measured.
* Urine or saliva will be collected to measure your nicotine, anabasine, and cotinine level.
* You will complete the same questionnaires you completed at the regular study visits.

This is an investigational study. Varenicline and the nicotine patch are both FDA approved and commercially available to help people stop smoking. The study doctor can explain how the study drugs are designed to work.

Up to 160 participants will be enrolled in this portion of the study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

Age: 18-75 years old

• Smoking 5 or more cigarettes, Little cigars and/or cigarillos per day, on average, within the 2 months preceding the screening visit and expired CO ≥ 6ppm (if ≤ 5, then NicAlert Strip >2).

* Interested in treatment that might change smoking behavior
* Able to follow verbal and written instructions in English and complete all aspects of the study
* Provide informed consent and agree to all assessments and study procedures
* Have an address and telephone number where they may be reached
* Be the only participant in their household

Exclusion Criteria:

Standard criteria for transdermal nicotine and varenicline smoking cessation trials will be used.

Exclusion criteria will include the following:

* Within the month immediately preceding the screening visit, use of any form of tobacco products other than cigarettes, little cigars and/or cigarillos on 3 or more days within a week if the individual refuses to refrain from such tobacco use during the course of the study.
* Current enrollment or plans to enroll in another smoking cessation program in the next 12 months
* Plan to use other nicotine substitutes (i.e., OTC or prescription medication for smoking cessation) or smoking cessation treatments in the next 12 months
* Uncontrolled hypertension (SBP greater than 180 or DBP greater than 110)
* Reports diagnosis of seizure disorder or a history of neurological illness or closed head injury that in the opinion of the PI feels that it would affect the results of the EEG
* History of severe kidney disease (e.g. chronic or acute kidney failure) with creatinine clearance below 30 and/or severe liver disease with liver tests over 4 times the upper normal level.
* Laboratory evaluations (kidney and liver) outside normal limits and of potential clinical significance in the opinion of the investigator
* Serious or unstable disease within the past 3 months
* History (last 3 months) of abnormal heart rhythms, cardiovascular disease (stroke, angina, heart attack) may result in ineligibility. These conditions will be evaluated on a case by case basis by the Study Physician.
* Current use of certain medications: (1) Smoking cessation meds (last 7 days), i.e., Wellbutrin, Bupropion, Zyban, NRT, Chantix, (2) Certain medications to treat depression (last 14 days), i.e.

MAOIs and Elavil (Amitriptyline), (3) A case by case determination will be made by study physician for medication on precautionary list, i.e. nitroglycerin, or (4) Daily use of opioids for 30 days or more on phone screen or at screening is exclusionary however PRN use is allowed (i.e., 3:7 days per week or less or if more frequent, use less than a month's duration.) --Meet criteria for the following psychiatric and/or substance use disorders as assessed by the MINI: items C (current manic or hypomanic episode only), I (alcohol abuse - Alcohol Addendum-past 6 months only; current alcohol dependence), J (substance abuse - Substance Abuse Addendum - past 6 months only; current substance dependence), K (current/lifetime psychotic disorder or current/lifetime mood disorder with psychotic features).

* Individuals who meet criteria for non-exclusionary psychiatric disorders that are considered clinically unstable and/or unsuitable to participate as determined by the Principal Investigator and/or Study Physician.

  * Individuals rated as moderate (9-16) to high (17 or greater) on suicidality as assessed by Module B of the MINI. --Psychiatric hospitalization within 1 year of screening date. --A positive urine pregnancy test during the screening period. Women who are two years postmenopausal, or who have had a tubal ligation or a partial or full hysterectomy will not be subject to a urine pregnancy test. --Pregnant, breast-feeding or of childbearing potential and is not protected by a medically acceptable, effective method of birth control while enrolled in the study. Medically acceptable contraceptives include: (1) approved hormonal contraceptives (such as birth control pills, patches, implants or injections), (2) barrier methods (such as a condom or diaphragm) used with a spermicide, or (3) an intrauterine device (IUD). Contraceptive measures sold for emergency use after unprotected sex are not acceptable methods for routine use. --History of hypersensitivity or allergic reaction to Varenicline, NRT, or any component of these formulations . --Any medical or psychiatric condition, illness, disorder, or concomitant medication that could compromise participant safety or treatment, as determined by the Principal Investigator and/or Study Physician.

    * Subject considered by the investigator as unsuitable candidate for receipt of an investigational drug, or unstable to be followed up throughout the entire duration of the study.
    * Positive toxicology screen for any of the following drugs: cocaine, opiates, methadone, benzodiazepines, barbiturates, amphetamines, methamphetamines, PCP, or THC.

      * A. Participants with valid prescriptions for opiates, benzodiazepines, barbiturates, amphetamines or methadone will not be excluded. B. Participants failing the toxicology screen will be allowed to re-screen once. If they test positive again, they will not be allowed to return.
    * Must not have visual problems that in the investigators opinion would interfere in the completion of the study assessments
    * Unwilling to change hairstyle or remove a wig as necessary for the appointment to accommodate the net that is required to be worn on the scalp during the study procedure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2015-12-14 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Continuous Nicotine Abstinence | 8 weeks
  Continuous abstinence over the last 4 weeks of treatment (i.e. EOT-end of treatment) will serve as the primary outcome measure. Saliva will be collected to measure cotinine level.

SECONDARY OUTCOMES:
Continuous and Prolonged Nicotine Abstinence | 3 months
  For prolonged abstinence, relapse defined by 7 or more consecutive days of smoking or smoking at least 1 cigarette over two consecutive weeks from the end of the grace period to a future time point (e.g., EOT, 3- and 6- months post-quit date).

CONTACTS AND LOCATIONS:
Overall Officials: Jason D Robinson, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org